CLINICAL TRIAL: NCT04315207
Title: Psychosocial Consequences of Receiving Results of Lung Cancer Workup by Telephone or In-person
Brief Title: Breaking Potentially Bad News in Lung Cancer Workup: Telephone Versus In-person Breaking of Final Diagnosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Naestved Hospital (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 12-000660
Record Dates: First submitted 2020-03-17; First posted 2020-03-19 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Lung Cancer; Diagnoses Disease; Psychosocial Stressor
Keywords: Invasive workup; Breaking bad news; Endoscopy
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized (1:1), controlled trial
Who Masked: Outcomes Assessor
Masking Description: Primary endpoint is a patient-reported outcome. Statistician were blinded to intervention until all statistical analyses were conducted
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- In-person visit (Active Comparator): In-person meeting with the patient in the out-patient department. The patient is free to bring up to four* relatives or other persons of their own choice to the in-person meeting.
  (* Restriction due to space limitation).
  Interventions: Behavioral: In-person meeting
- Telephone call (Experimental): Telephone call with the patient. The patient is free to turn on loudspeaker to include relatives or other persons in the telephone conversation, alternatively to ask the physician to call and inform one relative or other person after the patient-doctor telephone call
  Interventions: Behavioral: Telephone call

INTERVENTIONS:
Behavioral: Telephone call — All patients are informed that they will receive a telephone call between 08 AM and 5 PM on workdays, as soon as the results of invasive workup are available. This is expectedly 3 to 5 days after invasive workup. At the telephone call, patients are free to ask for a later call, to summon relatives, to turn on the loud speaker, and/or ask the physician to call one relative of choice to share the information.
  Regardless of group, all patients are informed on the possibility of malignancy at every patient-physician encounter.
  Arms: Telephone call
Behavioral: In-person meeting — All patients are provided a written and verbal appointment date 5 workdays after invasive workup, and that they will receive a telephone call if 1) results are not available at the time of the meeting, and/or 2) if results need urgent action (such as small-cell lung cancer).
  At the in-person meeting, patients are free to invite family and relatives (up to 4 persons, restriction due to space available).
  Regardless of group, all patients are informed on the possibility of malignancy at every patient-physician encounter.
  Arms: In-person visit

SUMMARY:
Disclosure of bad news is challenging for patients, relatives and healthcare providers. Current protocols for breaking bad news assume a single, in-person meeting for breaking bad news, however cancer workup is not a single event but a consecutive process with several contacts between patient and physician. Furthermore, an increasing number of patients receive their cancer diagnosis by telephone.

The investigators want to examine whether having the result of lung cancer workup by telephone results in worse psychosocial consequences than having the result in-person. Both groups receive information on possibility of cancer at every patient-physician contact.

DETAILED DESCRIPTION:
Lung cancer is the most common cause of cancer death worldwide. Patient-friendly delivery of results of lung cancer workup is mandatory in an era of personalized medicine. The possibility of delivering health care using telephone has been acknowledged for various medical interactions such as genetic counselling, delivery of screening results, smoking cessation programmes, palliative interventions, and disclosing result of breast cancer workup. However, Retrospective observational studies have identified higher patients' satisfaction scores when the cancer diagnosis is conveyed by a physician with high communicative skills, in personal rather than in impersonal settings, in-person rather than by telephone, when the patients had a perception of opportunity to ask questions, and when conversations lasted more than10 minutes and included discussion of treatment options.

All current models for breaking bad news (SPIKES, Kayes' 10 step-model, PACIENTE, BREAK) all focus on a single patient-physician encounter, which is in contrast to the organization of contemporary cancer workup as a flow of examinations and thus multiple encounters.

The study aims to examine the effects on psychosocial consequences of receiving the final diagnosis of workup of suspected cancer in lung, pleura or mediastinum by telephone versus in-person when patients receive information on possible malignancy at every patient-physician encounter.

HYPOTHESES:

The main hypothesis of this study is that having the final diagnosis of cancer workup delivered by telephone (intervention group) is associated with worse psychosocial consequences than when delivered in-person (control group). More specifically, the hypothesis is:

1) Receiving the result of cancer workup results in decreased scores of the disease-specific questionnaire Consequences of Screening: Lung Cancer (COS-LC) compared to patients receiving their results in-person.

Potential moderators and mediators:

During the study potential mediating and moderating factors will be explored, e.g. including socio-demography, comorbidity, and disease-specific factors, will be investigated. Most importantly, results on patients with confirmed cancer are explored separately as will data on patients without a final diagnosis of malignancy.

METHODS:

Study design:

The study is a non-pharmacological two-armed randomized controlled trial with intervention group receiving the result of cancer workup by telephone (telephone group) and active control group receiving result of cancer workup in-person ("gold standard"; in-person group). Both groups will otherwise receive the same information and in the same way, thus regardless of group, all patients are informed on the possibility of malignancy at every patient-physician encounter.

ELIGIBILITY:
Inclusion Criteria:

(all are mandatory)

1. suspicions lesions in lung, chest wall or mediastinum at CT or PET-CT
2. a clinician's decision of invasive work-up for suspected or possible malignancy.
3. expected survival of more than 5 weeks (as judged by a local investigator).

Exclusion Criteria:

1. age younger than 18 years
2. need of in-patient care
3. disease manifestation needing urgent care (e.g. spinal cord compression, superior vena cava superior syndrome) and
4. inability to provide verbal and written informed consent -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2012-10-01 (Actual); Primary Completion 2017-04-19 (Actual); Study Completion 2019-09-15 (Actual)

PRIMARY OUTCOMES:
Change in psychosocial consequences | Four weeks after receiving final diagnoses, equaling approximately 5 weeks randomization
  Questionnaire COS-LC (Consequences of Screening - Lung Cancer) part 1. COS-LC part 1 consists of nine psychosocial scales (four core and five lung-cancer-screening-specific scales). Each scale is constructed from an individual number of items (see below), and each item has four response categories ordered on a continuum: "not at all", "a bit", "quite a bit" and "a lot": The minimum score of each item is 0 with a maximum of 3. The higher the scale score, the more negative the psychosocial consequences The four core scales measure "Anxiety" (7 items; scale score 0-21), "Behaviour" (7 items; scale score 0-21), "Dejection" (6 items; scale score 0-18), and "Sleep" (4 items; scale score 0-12).
  The five lung-cancer-screening-specific scales measure "Self-blame" (5 items; scale score 0-15), "Focus on Airway Symptoms" (2 items; scale score 0-6), "Stigmatisation" (4 items; scale score 0-12), "Introvert" (4 items; scale score 0-12), and "Harm of Smoking" (2 items; scale score 0-6).

SECONDARY OUTCOMES:
Patient-perceived change at follow-up | Four weeks after receiving final diagnoses, equaling approximately 5 weeks randomization
  COS-LC part 2 encompasses six scales (24 items) focusing on patient-perceived changes at the time of follow-up (4 weeks after the final screening result) compared to baseline: "Calm/Relaxed" (2 items), "Social Relations" (3 items), "Existential Values" (6 items), "Impulsivity" (6 items), "Empathy" (3 items), and "Regretful of still Smoking" (4 items). All items in COS-LC part 2 have five response categories scored laterally reversed: "much less" 2, "less" 1, "the same as before" 0, "more" 1, and "much more" 2: Part 2 was designed and validated to measure changes, both positive and negative, and high scores denote more change

CONTACTS AND LOCATIONS:
Overall Officials: Uffe Bodtger, PhD, Principal Investigator — Dep. of Respiratory Medicine; Naestved Hospital; John Brodersen, PhD, Study Chair — University of Copenhagen
Locations (1):
- Department of Respiratory Medicine, Næstved, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Troubles concerning Danish data protection regulations in sharing outside Denmark